CLINICAL TRIAL: NCT05034198
Title: Development and Pilot Testing of a Remote Training Strategy for the Implementation of Mental Health Evidence-Based Practices in Rural Schools
Brief Title: Remote Training in Rural Schools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Devereux Center for Effective Schools (Unknown); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-017895; R18HS027755 (AHRQ)
Record Dates: First submitted 2021-09-01; First posted 2021-09-05 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Behavior Disorders
Keywords: Positive-behavior Interventions and Supports; Evidence-based Practices; Tier 2; Mental Health; Rural Schools
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being | interventions — Cognitive Behavioral Therapy; Schools

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stakeholder Input (No Intervention): Behavioral health staff (BHS) will be asked to complete two semi-structured qualitative interviews and a set of surveys. The first interview will be about perceived barriers and facilitators on utilizing a remote training platform. The second interview will cover perceived feasibility and acceptability of the proposed training, consultation, and the implementation of evidence-based practices. The surveys will ask about the perceived acceptability, appropriateness, and feasibility of the remote training platform.
- Asynchronous Training Development (No Intervention): Mental health trainers with expertise in the treatment of externalizing and internalizing behavior disorders will video-record the training modules and produce them using lecture capture technology (i.e., showing speaker and Power Point slides on a split screen). Each training module will be approximately 45 minutes long.
- Initial Mini-Tiral (Experimental): BHS will be given a procedures manual with instructions on how to access the video-recorded training modules on-demand. All participants will take part in this mini-trial. Immediately after BHS watch the videos, they will be asked to complete three brief surveys regarding the appropriateness, feasibility and acceptability of each training module and provide comments about each.
  Interventions: Behavioral: Coping Power Program (CPP); Behavioral: Cognitive behavioral therapy (CBT) for Anxiety Treatment in Schools (CATS); Behavioral: Check-in/Check-out (CI/CO)

INTERVENTIONS:
Behavioral: Coping Power Program (CPP) — CPP is an evidence-based intervention designed for students with externalizing behavior disorder. CPP consists of twelve 45-minute sessions. This EBP has been found to be effective at reducing aggressive behavior, covert delinquent behavior and substance abuse among aggressive boys, with gains maintained at one-year follow-up. Growth curve analyses showed that CPP had linear effects for three years after intervention on reductions in aggressive behavior and academic behavior problems.
  Arms: Initial Mini-Tiral
Behavioral: Cognitive behavioral therapy (CBT) for Anxiety Treatment in Schools (CATS) — CATS is an adaptation of Friends for Life (FRIENDS). The adapted protocol retains the core elements of evidence-based CBT for anxiety and the FRIENDS group format. Investigators implemented planned adaptations to the protocol based on collective experience. Changes were made to the language, cultural methods, number of sessions, and activities while maintaining the 5 essential components of the treatment. This resulted in a briefer (8-session) and more feasible, engaging and culturally appropriate protocol for urban under-resourced schools than the original FRIENDS.
  Arms: Initial Mini-Tiral
Behavioral: Check-in/Check-out (CI/CO) — CI/CO is a targeted, Tier 2 intervention for students at risk of developing externalizing and internalizing mental health disorders. CI/CO is designed to provide immediate feedback (i.e., at the end of each class period) to students, based on the use of a daily report card. This feedback is developmentally sensitive. CI/CO implementers meet individually with students for a brief 'check-in' in the morning and a brief 'check-out' in the afternoon. Research on the use of CI/CO has shown it to be effective in reducing externalizing and internalizing problems with elementary school students. CI/CO will be offered to individual students for a three-month period of time, which is the same time-frame needed for the implementation of CPP.
  Arms: Initial Mini-Tiral

SUMMARY:
Rural areas have fewer, and less well trained, health care providers than non-rural areas. Schools have become more involved in the delivery of mental health services and hold great potential for increasing access to children and adolescents. Innovations in training and service delivery are needed to improve mental health care quality and availability in rural schools. Evidence-based practices (EBPs) can be incorporated into school-wide multi-tiered systems that are currently used to improve school climate and safety. School-wide Positive Behavioral Interventions and Supports (PBIS), a service-delivery strategy based on the public health model is one example. Investigators will use an iterative process (Rapid Prototyping) to develop and evaluate the appropriateness, feasibility, acceptability, and preliminary efficacy of a remote training strategy that provides resources to support use of Tier 2 EBPs and effective support for care coordination practices in rural schools.

ELIGIBILITY:
Inclusion Criteria:

Any BHS (e.g., school counselor, school social worker or teacher who is under employment from a school district) based at a school implementing PBIS and who may be nominated by the principal as a potential participant is eligible to be included in the study. Additionally, the research staff will reach out to school behavioral health staff concurrently with the school principal. BHS staff will provide consent to participate.

Exclusion Criteria:

Staff from schools not implementing PBIS.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Stakeholder Input | Up to 2 years
  Semi-structured interviews and surveys will be conducted with stakeholders to determine efficacy of a universal strategies that provides resources to support evidence-based practices (EBPs) for implementing appropriate behavioral care coordination practices for students in rural schools in Pennsylvania.
Asynchronous Training Platform Development | Up to 2 years
  A Rapid prototyping approach will be used to develop non-interactive, remote training strategy (RTS) using on-demand, pre-recorded training videos for school personnel in rural schools based on preliminary studies and Aim 1 data.
Synchronous Training Platform Development | Up to 2 years
  A Rapid prototyping approach will be used to develop a remote training strategy (RTS) consisting of virtual meetings for school personnel in rural schools based on preliminary studies and Aim 1 data

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Eiraldi, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Eiraldi R, McCurdy BL, Khanna MS, Goldstein J, Comly R, Francisco J, Rutherford LE, Wilson T, Henson K, Farmer T, Jawad AF. Development and evaluation of a remote training strategy for the implementation of mental health evidence-based practices in rural schools: pilot study protocol. Pilot Feasibility Stud. 2022 Jun 17;8(1):128. doi: 10.1186/s40814-022-01082-4. PMID 35710520